CLINICAL TRIAL: NCT04255836
Title: A Pilot Study of Durvalumab Combined With Chemotherapy and Stereotactic Body Radiotherapy (SBRT) in Patients With Oligometastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: Durvalumab Combined With Chemotherapy and Stereotactic Body Radiotherapy (SBRT) in Patients With Oligometastatic Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-19-20392
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab therapy (Experimental): Chemo+Durvalumab (PD-L1 monoclonal antibody)1500 mg every 3 weeks [q3w] intravenously [iv] for 4 cycles, then SBRT 50-60 Gy/≤10f + Durvalumab 1500 mg q4w, then Durvalumab 1500 mg q4w for up to 24 months or until progression or other discontinuation criteria are met.
  Interventions: Drug: Durvalumab; Drug: the first line chemotherapy for metastatic NSCLC; Radiation: stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500mg q3w combined with chemotherapy for 4 cycles, then 1500mg q4w combined with SBRT, then 1500mg q4w for PD or up to 24 months
  Other Names: IMFINZI
Drug: the first line chemotherapy for metastatic NSCLC — paclitaxel+carboplatin or pemetrexed+cisplatin
Radiation: stereotactic body radiotherapy (SBRT) — SBRT total doses of 50-60Gy/≤10F

SUMMARY:
This is a Phase II, multi-center pilot study assessing the efficacy and safety of durvalumab combined with chemotherapy and stereotactic body radiotherapy (SBRT) in patients with oligo-metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer
* ≤3 metastatic organs and ≤5 metastatic lesions (supraclavicular and mediastinal lymph nodes are not classified as distant metastasis; other lymph node
* metastasis一group lymph node region will be classified as one metastatic lesion）
* Tissue biopsy prior to treatment
* ECOG performance score 0-1

Exclusion Criteria:

* EGFR mutation or ALK positive.
* Evidence on pulmonary interstitial disease or symptoms of active non-infectious pneumonia.
* Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus.
* Previous treatment with antibody against pd -1, pd - L1, pd - L2, CD137 or CTLA-4 (including ipilimumab or any antibody or drug against T cell co-stimulation or checkpoint pathway).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 2 years
  Progression-Free Survival (PFS) assessed according to RECIST 1.1 in subpopulation of patients with oligometastatic NSCLC

SECONDARY OUTCOMES:
Safety (AESI, AEs/SAEs) | up to 2 years
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
To assess the treat failure patterns | up to 2 years
  Treat failure patterns including local failure and distant metastasis
Objective response rate(ORR) | up to 2 years
  ORR was defined as the proportion of participants with partial response (PR) or complete response (CR) to treatment as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
and OS Overall Survival(OS) | up to 2 years
  OS was defined as the time from the date of enrollment until death by any cause. Participants still alive at the time of data analysis were censored at the date of last follow-up.